CLINICAL TRIAL: NCT02036736
Title: Randomized Study Evaluating the Influence of the Strategy Intraoperative Anesthetic (Desflurane Versus Propofol) on Cognitive and Psychomotor Functions in Output Post Interventional Room Monitoring
Brief Title: Evaluating the Influence of the Strategy Intraoperative Anesthetic (Desflurane Versus Propofol) on Cognitive and Psychomotor Functions in Output Post Interventional Room Monitoring - COGNIDES
Acronym: Cognides
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P120702; 2012-005270-61 (Other: eudraCTNumber)
Record Dates: First submitted 2014-01-08; First posted 2014-01-15 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2013-03

CONDITIONS: Orthopedic Surgery; Total Hip Prosthesis; Total Knee Replacement
Keywords: Orthopedic Surgery; Total hip prosthesis; Total knee replacement; Intraoperative anesthetic strategy; Propofol; Desflurane

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propofol (Experimental): Intraoperative anesthetic strategy by Propofol versus Desflurane
  Interventions: Drug: Intraoperative anesthetic strategy by Desflurane
- Desflurane (Experimental): Intraoperative anesthetic strategy by Desflurane versus Propofol
  Interventions: Drug: Intraoperative anesthetic strategy by Propofol

INTERVENTIONS:
Drug: Intraoperative anesthetic strategy by Propofol — 1- Arm Propofol: Propofol TCI induction target between 2 and 6 mg / mL
  * Sufentanil (0.15 mg / kg intravenously (IV))
  * Atracurium (0.5 mg / kg IV) Maintenance mode by Propofol TCI target between 2 and 4 micrograms / mL tune to 40 <BIS <60 Sufentanil bolus according to intraoperative analgesia Atracurium bolus according to the level of neuromuscular blockade
  Arms: Desflurane
Drug: Intraoperative anesthetic strategy by Desflurane — 2- Arm Desflurane Desflurane induction (2-3 mg / kg)
  * Sufentanil (0.15 mg / kg IV)
  * Atracurium (0.5 mg / kg IV)) Desflurane closed by maintenance target with minimal alveolar concentration (MAC) to adapt the circuit to obtain a figure 40 <BIS <60 Sufentanil bolus according to intraoperative analgesia Atracurium bolus according to the level of neuromuscular blockade
  Arms: Propofol

SUMMARY:
The recovery of cognitive and psychomotor functions is best performed under anesthesia after desflurane when propofol in that obtaining a Aldrete score> 8/10 output of the allowing SSPI.

The principal objective is to compare the cognitive and psychomotor status of patients recovered an Aldrete score> 8/10 according to the anesthetic agent (propofol or desflurane) using three tests (Stroop test, Digit Symbol Substitution task and a test of verbal memory (visual verbal learning test) made SSPI.

DETAILED DESCRIPTION:
The day before surgery, patients sign the consent and will be randomized. Then 3 tests (Stroop test, Digit Symbol Substitution Task and visual verbal learning test) will be performed. No anxiolysis will be given to the patient. The anesthetic induction will be with IV propofol (2-3 mg / kg). The maintenance will anesthetic, desflurane by for a minimum alveolar concentration of between 2% and 6% or propofol for intravenous anesthesia user target controlled. In SSPI, the Aldrete score will be evaluated every 5min. Upon obtaining a Aldrete score> 8/10, the day before the tests will be carried out again

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 80 years
* ASA I, II
* General anesthesia provided
* Scheduled orthopedic surgery
* Duration of surgery between one and three hours
* Patient has given its written consent
* Patient receiving medical health insurance

Exclusion Criteria:

* MMS (Mini Mental State) ≤ 24
* Patient does not speak or read or do not understand the French
* Previous surgery within seven days
* Coronary insufficiency, renal, hepatic
* Chronic pulmonary disease
* Obesity (BMI> 35)
* Addiction
* Chronic alcoholism
* Hematocrit <25%
* Personal and family history of malignant hyperthermia
* Taking benzodiazepines or psychotropic within 24 hours preoperative
* Psychiatric pathology being
* Psychological or neurological disorder causing difficulties in understanding the study
* Chronic pain and / or taking analgesics 3.
* Pregnancy or breastfeeding
* Disorder of hemostasis: platelets <80,000 / mm3, PT <50% TCA> 1.5 times the control.
* Hypersensitivity to propofol or desflurane or any of the excipients
* Patients allergic to soy and peanuts
* History of liver disease, jaundice, unexplained fever, eosinophilia after administration of a halogenated anesthetic
* Hypersensitivity to egg lecithin.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Compare the cognitive and psychomotor status of patients recovered an Aldrete score> 8/10 according to the anesthetic agent (propofol or desflurane) | 1 day
  Compare the cognitive and psychomotor status of patients recovered an Aldrete score> 8/10 according to the anesthetic agent (propofol or desflurane), using three tests (Stroop test, Digit Symbol Substitution Task and test verbal memory (visual verbal learning test) made room post-interventional monitoring
  The primary endpoint will be the average score of three tests in room post-interventional monitoring (Stroop test, Digit Symbol Substitution Task, Visual Verbal Learning Test) scores expressed in standard deviation

SECONDARY OUTCOMES:
proportion of patients with nausea and vomiting | 1 day
Search intraoperative factors alterations in cognitive and psychomotor functions (number of red blood cells transfused, number of hypotensive episodes (≤ 80mmHg or MAP NOT ≤ 65mmHg)≥ 10 minutes). | 1 day
Evaluate patient satisfaction on a visual analogue scale in room post-interventional monitoring | 1 day
Evaluate postoperative pain in room post-interventional monitoring | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Cyrille Robert, PH, Principal Investigator — APHP
Locations (1):
- Hôpital Saint Antoine, Paris, Paris, France